CLINICAL TRIAL: NCT02700529
Title: Ubenimex in Adult Patients With Lymphedema of The Lower Limb: a Phase 2, RAndomized, Double-blind, Placebo-controlled Study of Efficacy, Safety, and Pharmacokinetics (ULTRA)
Brief Title: Ubenimex in Adult Patients With Lymphedema of The Lower Limb (ULTRA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EIG-UBX-003
Record Dates: First submitted 2016-02-26; First posted 2016-03-07 (Estimated); Results first posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — ubenimex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- ubenimex (Experimental): ubenimex capsules 150 mg three times a day (TID), administered orally for a total of 24 weeks.
  Interventions: Drug: ubenimex
- placebo (Placebo Comparator): matched placebo capsules TID, administered orally for a total of 24 weeks
  Interventions: Other: placebo

INTERVENTIONS:
Drug: ubenimex
  Other Names: UBX
  Arms: ubenimex
Other: placebo
  Arms: placebo

SUMMARY:
This proof-of-concept study is designed as a randomized, double-blind, placebo-controlled study comparing ubenimex at 150 mg, 3 times daily (total daily dose of 450 mg) with placebo for 6 months treatment period in patients with leg lymphedema.

DETAILED DESCRIPTION:
Leukotriene B4 (LTB4) inhibits lymphangiogenesis in the mouse tail model of lymphedema and is elevated in tissue in patients with lymphedema. Ubenimex is an inhibitor of leukotriene A4 hydrolase (LTA4H), the biosynthetic enzyme for LTB4. This proof-of-concept study is designed as a randomized, double-blind, placebo-controlled study comparing ubenimex at 150 mg, 3 times daily (total daily dose of 450 mg) with placebo for 6 months treatment period in patients with leg lymphedema. The primary objectives for the study are:

* To evaluate the efficacy of ubenimex in patients with leg lymphedema
* To evaluate the safety and tolerability of ubenimex in patients with leg lymphedema

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of secondary leg lymphedema, based on a positive lymphoscintigraphy (LSG) study of the affected leg OR has a diagnosis of primary lymphedema not of congenital onset affecting one or both lower limbs, based on positive LSG.
2. Swelling of at least 1 leg not completely reversed by leg elevation or compression.
3. Stage II or greater lymphedema, based on the International Society of Lymphology (ISL) staging system.
4. Completion of a full course of complete decongestive therapy (CDT).
5. Stable limb volume (within 10% during screening for worse/affected leg) .
6. If patient has had a lymphatic vascularization procedure (lymphovenous bypass or lymph node transfer) or liposuction for lymphedema in the affected limb, then procedure must have been performed at least 1 year (12 months) prior to Screening AND affected limb must be clinically stable over the 3 months prior to Screening AND significant residual disease must be present.
7. Ambulatory status (use of a walking aid is permitted).
8. Agree to use a medically acceptable method of contraception, if the possibility of conception exists.

Exclusion Criteria:

Exclusions Based on Lymphedema:

1. A diagnosis of primary lymphedema with congenital onset. Primary lymphedema is defined as lymphedema with onset prior to or without an inciting event (e.g, surgery, trauma, radiation)
2. Occurrence of significant lymphedema of another body part that is not the lower limb (e.g, upper extremity, trunk, head and neck, genitalia).
3. Lymphedema involving all four limbs
4. Recent initiation of, or intention to initiate CDT or maintenance physiotherapy for lymphedema.

   Exclusions Based on Other Medical Conditions
5. Deep venous thrombosis in either lower limb or systemic anticoagulation within 6 months
6. Other medical condition that could lead to acute or chronic leg edema.
7. Other medical condition that could result in symptoms overlapping those of lymphedema in the affected leg.
8. History of clotting disorder (hypercoagulable state).
9. Chronic (persistent) infection in either lower limb.
10. Cellulitis or other infection in either lower limb or use of antibiotics for cellulitis within 3 months prior to screening.
11. Other unstable or severe medical condition requiring active management and/or likely to decompensate/require active management within the next year
12. Current evidence of malignancy.
13. History of malignancy within the previous 3 years, except for nonmelanoma skin cancer or cervical carcinoma in situ treated with curative intent.
14. Currently receiving chemotherapy or radiation therapy.
15. Life expectancy < 2 years for any reason.
16. Pregnancy or nursing.
17. Substance abuse (such as alcohol or drug abuse) within 6 months prior to screening.

    Exclusions Based on Concurrent Medication Use
18. Regular concurrent use or regular use within 6 months before screening of another leukotriene pathway inhibitor.
19. Concurrent antibiotic use.
20. Concurrent use of any agent active on the sphingosine-1-phosphate (S1P) pathway.
21. Concurrent use of unapproved (including herbal) treatments for lymphedema.

    Exclusions Based on Laboratory Values
22. Significant or chronic renal insufficiency or requires dialytic support.
23. Hepatic dysfunction.
24. Absolute neutrophil count <1500 mm3 at screening.
25. Hemoglobin concentration <9 g/dL at screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-06; Primary Completion 2018-10 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Stanford University, Stanford, California
  - Orlando Health, Inc., Orlando, Florida
  - The Ohio State University Wexner Medical Center James Cancer Hospital, Columbus, Ohio
- Macquarie University Hospital (MUH), Sydney, New South Wales, Australia

REFERENCES:
- [Background] Orning L, Krivi G, Fitzpatrick FA. Leukotriene A4 hydrolase. Inhibition by bestatin and intrinsic aminopeptidase activity establish its functional resemblance to metallohydrolase enzymes. J Biol Chem. 1991 Jan 25;266(3):1375-8. PMID 1846352

RESULTS

PARTICIPANT FLOW:
Groups:
- Ubenimex: ubenimex capsules 150 mg three times a day (TID), administered orally for a total of 24 weeks.
  ubenimex
- Placebo: matched placebo capsules TID, administered orally for a total of 24 weeks
  placebo
Period: Overall Study
Arm/Group | Ubenimex | Placebo
Started | 27 | 27
Completed | 26 | 27
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ubenimex | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Full Range); unit: years] | 55.0 [38 to 74] | 53.4 [23 to 73] | 54.2 [23 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 0 | 2
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Type of Lymphedema [Count of Participants; unit: Participants]
  Secondary Lymphedema | 21 | 18 | 39
  Primary Lymphedema | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Skin Thickness of the Calf of the Most Affected Leg, Measured by Skinfold Calipers
Description: Change from baseline to Week 24 in skin thickness of the calf of the most affected leg, measured by skinfold calipers in the Skin-Thickness Intent-to-Treat (ST-ITT) population (patients with skin thickness >/= 10 mm at baseline) which comprised of 36 patients (16 ubenimex, 20 placebo).
Time Frame: Baseline through Week 24
Population: ST-ITT population (patients with skin thickness >/= 10 mm at baseline) which comprised of 36 patients (16 ubenimex, 20 placebo)
Measure: Mean (Standard Error); unit: mm
Arm/Group | Ubenimex | Placebo
Number analyzed (Participants) | 16 | 20
mm | -6.83 (1.913) | -7.75 (1.657)

ADVERSE EVENTS:
Time Frame: 7 months
Groups:
- Ubenimex: ubenimex capsules 150 mg three TID, administered orally for a total of 24 weeks.
  ubenimex
Arm/Group | Ubenimex | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/27 | 1/27
Other Adverse Events (participants affected / at risk) | 13/27 | 4/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ubenimex (N=27) | Placebo (N=27)
Supraventricular tachycardia / (Cardiac disorders) | 1 | 0
Adnexal torsion (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ubenimex (N=27) | Placebo (N=27)
Headache (Nervous system disorders) | 4 | 4
Feeling abnormal (Nervous system disorders) | 3 | 0
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 | 0
vomiting (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/29/NCT02700529/Prot_SAP_000.pdf